CLINICAL TRIAL: NCT02633813
Title: A Randomized, Prospective Multicenter, Double Blind, Parallel Assignment Placebo Controlled BE Study Of Naftifine Hydrochloride 2% Topical Cream With Naftin® In Patients With Tinea Pedis Using Clinical Endpoints
Brief Title: BE Study of Naftifine HCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzum Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-13-661
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Tinea Pedis
Keywords: Bioequivalence; Tinea pedis; Naftin
MeSH Terms: conditions — Tinea Pedis | interventions — naftifine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naftifine hydrochloride 2% (Experimental): A thin layer of sufficient quantity of Naftifine hydrochloride cream need to be applied to the affected areas plus an approximate ½ inch margin of healthy surrounding skin once daily consecutively for 2 weeks.
  Interventions: Drug: Naftifine hydrochloride 2%
- Naftin® 2% (Naftifine hydrochloride 2%) (Active Comparator): A thin layer of sufficient quantity of Naftifine hydrochloride cream need to be applied to the affected areas plus an approximate ½ inch margin of healthy surrounding skin once daily consecutively for 2 weeks.
  Interventions: Drug: Naftin® 2% (Naftifine hydrochloride 2%)
- Placebo vehicle cream. (Placebo Comparator): A thin layer of sufficient quantity of vehicle cream need to be applied to the affected areas plus an approximate ½ inch margin of healthy surrounding skin once daily consecutively for 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naftifine hydrochloride 2% — Topical application for two weeks
  Other Names: Naftifine hcl
  Arms: Naftifine hydrochloride 2%
Drug: Placebo — Topical application for two weeks
  Other Names: Vehicle cream
  Arms: Placebo vehicle cream.
Drug: Naftin® 2% (Naftifine hydrochloride 2%) — Topical application for two weeks
  Other Names: Naftifine hcl
  Arms: Naftin® 2% (Naftifine hydrochloride 2%)

SUMMARY:
The current study was randomized, double blind, placebo-controlled, prospective, multicenter, comparative therapeutic equivalence study.

The study duration for each patient was 6 weeks: Following were the visit details.

V1-Baseline and Randomization Visit (Day 1). V2- End of therapy visit (at the end of week 2 + 2 days). V3- Follow up visit (at the end of week 4 + 2 days). V4 - Test of cure visit ( at the end of week 6 + 4 days).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females aged more than or equal to 18 years
2. Clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot (the non-interdigital lesions should not be hyperkeratotic, i.e., characteristic of tinea pedis moccasin), and provisionally confirmed at baseline by a positive potassium hydroxide (KOH) wet mount preparation (i.e., skin scrapings from the target site are placed on a microscope slide with a drop of 10% KOH, and microscopic examination reveals segmented fungal hyphae)
3. The sum of the clinical signs and symptoms scores of the target lesion is at least 4, including a minimum score of at least 2 for erythema AND a minimum score of 2 for either scaling or pruritus (on a scale of 0-3, where 2 indicates moderate severity)

Exclusion Criteria:

1. Pregnant or lactating or planning to become pregnant during the study period
2. Use of antipruritics, including antihistamines, within 72 hours prior to entry into the study
3. Use of topical corticosteroid, antibiotics or antifungal therapy within 2 weeks prior to entry into the study
4. Use of systemic (e.g., oral or injectable) corticosteroid, antibiotics or antifungal therapy within 1 month prior to entry into the study
5. Use of oral terbinafine or itraconazole within 2 months prior to entry into the study
6. Use of immunosuppressive medication or radiation therapy within 3 months prior to entry into the study.
7. Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface.
8. Presence of any other infection of the foot or other disease process that might confound the treatment evaluation
9. History of dermatophyte infections unresponsive to systemic or topical antifungal drugs
10. Known hypersensitivity to Naftifine Hydrochloride or to any component of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mycological cure and clinical cure for a single target lesion for Trichyphyton rubrum | week 6 + 4 days
  After 6 weeks the skin scrapping will be collected for culture to find out the growth of T rubrum. Absence of growth suggests complete cure.

SECONDARY OUTCOMES:
Mycological cure and clinical cure for Trichophyton rubrum, Trichophyton mentagrophytes, or Epidermophyton floccosum | week 6 + 4 days
  After 6 weeks the skin scrapping will be collected for culture to find out the growth of T rubrum, T Mentagrophytes or E floccosum. Absence of growth suggests complete cure.

OTHER OUTCOMES:
Assessment of AEs for each treatment groups | week 6 + 4 days
  number of adverse events reported will be collated from all the treatment arms, to evaluate the safety of the study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Zaidoon Al-Zubaidy, Study Chair — Catawba Research
Locations (14):
- United States (12):
  - Moore Clinical Research Inc, Brandon, Florida
  - Savin Medical Group Research, Miami, Florida
  - International Dermatology Research, Inc,, Miami, Florida
  - FXM Research Corp, Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - South Tampa, MOORE Clinical Research, Inc., Tampa, Florida
  - North Tampa MOORE Clinical Research, Inc., Tampa, Florida
  - Medi Search, Saint Joseph, Missouri
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Research Across America, Dallas, Texas
  - Family Practise, Mesquite, Texas
  - Research Across America, Plano, Texas
- Dominican Republic (2):
  - Instituto Dermatológico y Cirugía de Piel, Santo Domingo, San Cristóbal
  - Instituto Dermatológico, Barrio Maria Auxiliadora, Santo Domingo Province

IPD SHARING:
Plan to Share IPD: Undecided